CLINICAL TRIAL: NCT03545490
Title: A Prospective, Randomized, Clinical Study to Evaluate the Effects of Early Enteral Nutritional Supplementation on Clinical Outcomes in Patients With Oral and Oropharyngeal Cancer Undergoing Radio(Chemo)Therapy After Surgical Resection
Brief Title: Early Enteral Nutritional Supplementation on Patients With Oral and Oropharyngeal Cancer Undergoing Radio(Chemo)Therapy After Surgical
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, Director, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANCH 1601
Record Dates: First submitted 2018-03-21; First posted 2018-06-04 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2020-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Cohort 1: nutritional supplements are given through oral route Cohort 2: nutritional supplements are given by tube feeding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1-intervention (Experimental): Oral supplements are given through oral route 2 weeks before radiotherapy.
  Interventions: Dietary Supplement: Early nutritional intervention
- Cohort 1-Control (Active Comparator): Oral supplements are given through oral route on demand during radiotherapy.
  Interventions: Dietary Supplement: Early nutritional intervention
- Cohort 2- Intervention (Experimental): Oral supplements are given by tube feeding 2 weeks before radiotherapy.
  Interventions: Dietary Supplement: Early nutritional intervention
- Cohort 2- Control (Active Comparator): Oral supplements are given by tube feeding on demand during radiotherapy.
  Interventions: Dietary Supplement: Early nutritional intervention

INTERVENTIONS:
Dietary Supplement: Early nutritional intervention — Early nutritional intervention (Ensure) was given two weeks before radiotherapy. Ensure 3 times per day, Mixing 55.8 g or 6 spoons of Ensure with 190 mL of warm water.

SUMMARY:
The target population in the present study is Chinese patients with oral and oropharyngeal cancer who plan to receive radio(chemo)therapy after surgical resection in the outpatient department. Investigators hypothesize that early enteral nutrition intervention, which is initiated 2 weeks before the start of postoperative radio(chemo)therapy treatment and added on demand during radiotherapy, will improve patients' nutritional status, tolerability to the radio(chemo)therapy, quality of life, and other clinical outcomes compared to commencement of oral nutritional supplements during the course of irradiation treatment. There are two cohorts in this trial, cohort 1 included patients with oral nutritional supplements and cohort 2 included patients with tube feeding (nasogastric tube or percutaneous endoscopic gastrostomy).

DETAILED DESCRIPTION:
This clinical trial will be conducted in a single-center, prospective, and randomized manner. In this protocol, the standard radio(chemo)therapy duration is 6-7 weeks. Early enteral nutrition intervention (EEN) refers to starting enteral nutrition intervention 2 weeks before post-operative radio(chemo)therapy begins and stopping this intervention when post-operative radio(chemo)therapy completes. Standard enteral nutrition intervention (SEN) refers to starting of enteral nutrition intervention on demand during (chemo)radiotherapy. Nutritional supplementation was given either through the oral route (Cohort 1) or tube feeding (nasogastric tube or percutaneous endoscopic gastrostomy, cohort 2). Dietitians will design meal plans for both groups of subjects so that their normal diets will provide 25-30 kcal/d/kg body weight in addition to nutritional supplements.

ELIGIBILITY:
Inclusion criteria

* Subject is male or female, between 18 and 70 years old;
* Subject has clinical or radiological diagnosis of oral cancer (stage III and stage IV), had surgical resection 3 or 4 weeks prior to radio (chemo)therapy, and plans to receive radio (chemo)therapy treatment;
* Subject has Karnofsky Performance Score (KPS) ≥ 60 and an expected life expectancy ≥ 6 months;
* Subject is willing to comply with the study protocol, able and willing to consume study product according to the protocol;
* Subject has voluntarily signed and dated the informed consent form (ICF), approved by an Institutional Review Board (IRB) / Independent Ethics Committee (IEC) prior to any participation in the study

Exclusion criteria

* Except for oral cancer and oropharyngeal cancer, subject has malignant tumors or serious infectious diseases, such as tuberculosis activity, respiratory system, cardiovascular system, urinary system diseases, systemic edema and ascites caused by diseases, etc., cannot participant in study in the opinion of study physician.
* Subject has dysfunction of liver, kidney or gallbladder, cannot participant in study in the opinion of study physician.
* Subject has gastrointestinal diseases to cannot tolerate enteral nutrition (such as intestinal bleeding, intestinal obstruction, severe digestive malabsorption, severe nausea and vomiting and diarrhea) that preclude his or her participation in the opinion of study physician;
* Subject has diabetes
* Subject has known history of allergy or intolerance to any ingredient in the investigational product;
* Female subjects are pregnant or plan to get pregnant within a year or are postpartum and non-lactating;
* Subject has mental illness, cannot understand ICF, unwilling to provide informed consent.
* Subject has amputation or implanted electronic devices or metal, it may be inappropriate to use BIA to measure body composition
* Subject is currently or has participated in any clinical trial 2 months prior to enrollment.
* Subject plans to take nutritional supplements and/or traditional Chinese medicine regularly during study in the opinion of study physician. Multi-vitamin and multi-mineral supplements are exception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 10 weeks
  changes of body weight from baseline to Final Visit/Exit.

SECONDARY OUTCOMES:
Body weight | 2weeks,5 weeks, 8 weeks
  Changes of body weight from baseline to V2, V3 and V4
Body Mass Index | 10 weeks
  Body Mass Index variables at baseline to V2, V3,V4 and Final Visit/Exit
Calf circumference by measure | 5weeks, 10 weeks
  Calf circumference variables at baseline to V3 and Final Visit/Exit
Lean mass measured by Bioelectrical impedance analysis (BIA) | 5weeks 10 weeks
  Lean mass variables at baseline, V3 and Final Visit/Exit
Fat mass measured by Bioelectrical impedance analysis (BIA) | 5weeks 10 weeks
  Fat mass variables at baseline, V3 and Final Visit/Exit
Patient-Generated Subjective Global Assessment/PG-SGA scores | 5weeks 10 weeks
  PG-SGA scores, an assessment tool for nutritional status at baseline, V3 and Final Visit/Exit.
  The Scored PG-SGA includes the four patient-generated historical components (Weight History, Food Intake, Symptoms and Activities and Function), the professional part (Diagnosis, Age, Metabolic stress, and Physical Exam), the Global Assessment (A = well nourished, B = moderately malnourished or suspected malnutrition, C = severely malnourished), the total numerical score, and nutritional triage Recommendations (0-1=No intervention required, 2-3 Education and lab values as appropriate, 4-8 Required intervention, >=9 Indicates a critical need for improved and/or nutrient intervention).
  Subtotal 4 historical components: scoring 0-30+
  * Weight history and Symptoms scores are additive
  * Food intake and Activities and Function, the highest point score,
  Professional component:
  * Criteria for condition, scoring 0-6
  * Metabolic Stress, scoring 0-3
  * Physical components, scoring 0-3
Dietary adherence and intake assessment | 2weeks,5 weeks, 8 weeks, 10 weeks
  Dietary adherence and intake assessment will be conducted by dietitians at V2, V3, V4 and Final Visit/Exit. Dietary adherence will be determined through comparing subjects' meal plans and actual consumptions as reflected by food diaries.
Prealbumin by drawing blood | 5weeks 10 weeks
  Prealbumin variables at baseline, V3 and Final Visit/Exit
Albumin by drawing blood | 5weeks 10 weeks
  Albumin variables at baseline, V3 and Final Visit/Exit
Hemoglobin by drawing blood | 5weeks 10 weeks
  Hemoglobin variables at baseline, V3 and Final Visit/Exit
White blood cell by drawing blood | 5weeks 10 weeks
  White blood cell variables at baseline, V3 and Final Visit/Exit
Peripheral blood lymphocyte by drawing blood | 5weeks 10 weeks
  Peripheral blood lymphocyte variables at baseline, V3 and Final Visit/Exit
Tolerability to radio(chemo)therapy assessment on treatment status | 5 weeks, 8 weeks, 10 weeks
  Treatment status (e.g., treatment course and doses completed as planned or changed) since last visit at V3, V4 and Final Visit/Exit
Tolerability to radio(chemo)therapy assessment on treatment change due to side effects | 5 weeks, 8 weeks, 10 weeks
  Number of days when treatment is suspended due to side effects since last visit at V3, V4 and Final Visit/Exit
Tolerability to radio(chemo)therapy assessment on complications | 5 weeks, 8 weeks, 10 weeks
  Incidence of radio(chemo)therapy-related complications such as oral mucositis, pneumonia, and shingles since last visit at V3, V4 and Final Visit/Exit
Tolerability to radio(chemo)therapy assessment on staying in hospital due to complications | 5 weeks, 8 weeks, 10 weeks
  Number of days when patients stay in hospital for treatment of radio(chemo)therapy-related complications since last visit at V3, V4 and Final Visit/Exit (if applicable)
Quality of life assessed by Quality of Life Questionnaire-Core 36 of European Organization for Research on Treatment of Cancer/EORTC Quality of Life QLQ-C30 questionnaire | 5 weeks, 8 weeks, 10 weeks
  Subjective assessment of physical activity, mood, fatigue and eating status by EORTC Quality of Life QLQ-C30 questionnaire at baseline, V3, V4 and Final Visit/Exit
Quality of life assessed by Quality of Life Questionnaire-Head and Neck 35 questionnaire of European Organization for Research on Treatment of Cancer/EORTC Quality of Life QLQ-H&N35 | 5 weeks, 8 weeks, 10 weeks
  Subjective assessment of physical activity, mood, fatigue and eating status by EORTC Quality of Life QLQ-H&N35 questionnaire at baseline, V3, V4 and Final
Health economics assessment on medications treatment due to complications | 10 weeks
  Costs for medications treated for radio(chemo)therapy-related complications during this study
Radio(chemo)therapy treatment effect | 10 weeks
  The variable is local tumor control probability assessed at baseline and Final Visit/Exit.
  Local tumor control probability is defined as the percentage of patients who do not have tumor recurrence in the total patients.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, Study Director — Shanghai 9th people hospital
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jiang W, Zhang H, Dou S, He Y, Zhu G, Li R. Effectiveness of Early Oral Nutritional Supplementation in Preventing Weight Loss in Head and Neck Cancer Patients Undergoing Postoperative Radiotherapy or Chemoradiotherapy: A Prospective Randomized Controlled Trial. J Am Nutr Assoc. 2025 Aug;44(6):498-507. doi: 10.1080/27697061.2025.2458277. Epub 2025 Feb 4. PMID 39903480